CLINICAL TRIAL: NCT02908633
Title: Comparison of Safety and Efficacy of Three Variants of Canaloplasty: Ab-externo, Ab-interno and Minicanaloplasty Combined With Phacoemulsification to Treat Glaucoma and Cataract. A Randomised, Prospective Study.
Brief Title: Safety and Efficacy of Three Variants of Canaloplasty With Phacoemulsification to Treat Glaucoma and Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Marek Rekas, MD, PhD Professor of Ophthalmology, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 76/WIM/2015; 76/WIM/015 (Other: MMI)
Record Dates: First submitted 2016-09-17; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Primary Open Angle Glaucoma, Cataract
Keywords: open angle glaucoma; canaloplasty; migs; abic
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- canaloplasty ab externo and phacoemulsification (Active Comparator): As soon as the two scleral flaps: deep and superficial -similar to deep sclerectomy are dissected, the phacoemulsification with PCIOL insertion is performed. After excision of the deep flap the descemets window and ostia of Schlemm canal are created, the microcatheter is placed in the canal and guided for 360 degrees within the canal. Surgeon observes the location of beacon tip through sclera and injects the Healon GV. Then a suture is tied to the distal tip and the microcatheter is withdrawn. As it appears at the other ostium of canal the microcatheter it separated from the suture.Then suture loop is tightened to tension the trabecular meshwork. The superficial flap is sutured watertight to prevent bleb formation
  Interventions: Procedure: canaloplasty and phacoemulsification
- canaloplasty ab interno and phacoemulsification (Active Comparator): This variant of canaloplasty spares conjunctival surface. First phacoemulsification and PCIOL placement is performed. The Schlemm's canal is reached through goniotomy through anterior chamber. Similarly microcatheter is inserted and viscodilatator applicated. The key difference, is that no tensioning suture is left after the catheter is withdrawn. phacoemulsification is performed.
  Interventions: Procedure: canaloplasty and phacoemulsification
- minicanaloplasty and phacoemulsification (Active Comparator): The dissected conjunctival flap is of minimal size. The scleral flaps are sized: superficial flap 3x1mm, and deep flap: 1x1 mm- with no removal of the deep flap. Afterwards phacoemulsification part is performed. The microcatheterization and viscodilatation are conducted as in the traditional procedure.The conjunctiva is closed with one suture or coagulation
  Interventions: Procedure: canaloplasty and phacoemulsification

INTERVENTIONS:
Procedure: canaloplasty and phacoemulsification
  Other Names: canaloplasty ab externo; canaloplasty ab interno; minicanaloplasty

SUMMARY:
It is a comparative study of Safety and Efficacy of Three Variants of Canaloplasty: ab-externo, ab-interno and minicanaloplasty. Combined With Phacoemulsification to Treat Glaucoma and Cataract. It is a Randomised, Prospective Study.

ELIGIBILITY:
Inclusion Criteria:

* co-existing glaucoma and cataract
* glaucoma types: primary open angle glaucoma,
* eye with characteristic glaucoma changes (biomicroscopic,visual field)
* IOP over 21 mmHg after washout
* patients not tolerating antiglaucoma medications,
* patients with poor compliance
* progression in visual field

Exclusion Criteria:

* previous surgical glaucoma procedure
* previous cataract surgery
* BCVA under 0,004
* closed angle glaucoma secondary glaucoma (pseudoexfoliative, pigmentary)
* poorly controlled diabetes mellitus
* advanced AMD
* active inflammatory disease
* pregnancy
* mental disease or emotional instability general steroid therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
mean IOP | change form baseline at 24 months
Number of antiglaucoma drugs | change from baseline at 24 months
intraoperative complications | at the day of surgery

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity | change from baseline at 24 months
Visual Field changes | change from baseline at 24 months
  MD,
Early and Late postsurgical complications | within 24 months
% IOP reduction | change at 24 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Poland

REFERENCES:
- [Derived] Danielewska ME, Kicinska AK, Placek MM, Lewczuk K, Rekas M. Changes in spectral parameters of corneal pulse following canaloplasty. Graefes Arch Clin Exp Ophthalmol. 2019 Nov;257(11):2449-2459. doi: 10.1007/s00417-019-04433-9. Epub 2019 Aug 3. PMID 31377849